CLINICAL TRIAL: NCT01563432
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of Febuxostat Between TMX-67 40mg 2 Tablets and Feburic® 80mg 1 Tablet in Healthy Male Volunteers
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Characteristics Between TMX-67 and Feburic® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TMX-67_BE_I_2011
Record Dates: First submitted 2012-03-16; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-02

CONDITIONS: Gout
Keywords: crossover; pharmacokinetic; hyperuricemia; gout
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- febuxostat (TR) (Experimental)
  Interventions: Drug: Feburic®; Drug: TMX-67
- febuxostat (RT) (Experimental)
  Interventions: Drug: Feburic®; Drug: TMX-67

INTERVENTIONS:
Drug: Feburic® — 80 mg*1 tablet
Drug: TMX-67 — 40 mg*2 tablets

SUMMARY:
This study was designed to compare and evaluate the pharmacokinetic characteristics of febuxostat after single oral administration of TMX-67 (test drug) and Feburic® tablet in healthy adults; and to evaluate safety and tolerance following a single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 20 and 45 years
* Subjects whose weight is 50 kg or more and BMI is between 18 and 29 kg/m2
* Subjects who were voluntarily decided to participate in the study and provided written informed consent to observe the directions

Exclusion Criteria:

* Medical history which may influence adsorption, distribution, metabolism, excretion of the drug
* Clinically significant active chronic disease(s)
* Persons who are deemed ineligible for the study by the investigator according to the clinical laboratory test results or for other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics (AUClast and Cmax) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 14, 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea